CLINICAL TRIAL: NCT03171792
Title: Experience of Chronic (Non-malignant) Musculoskeletal Pain of French Adolescent and Young Adult: a Qualitative Research With Their Physicians and Non-medical Practitioners
Acronym: DMS-AJA
Status: Completed | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: URC-CIC Paris Descartes Necker Cochin (Other)
Responsible Party: Sponsor
Other Study IDs: NI16015; 2017-A00842-51 (Other: ANSM)
Record Dates: First submitted 2017-05-26; First posted 2017-05-31 (Actual); Last update posted 2025-11-20 (Actual); Status verified 2025-09

CONDITIONS: Chronic (Non-malignant) Musculoskeletal Pain
Keywords: Musculoskeletal pain; Adolescent; Qualitative research; Attitude; Health professionals
MeSH Terms: conditions — Bronchiolitis Obliterans Syndrome; Musculoskeletal Pain; Behavior

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: semi-structured interviews — Semi-structured face to face or telephone interviews with an open-ended approach. Duration: about 45 minutes. Audio-recorded. Exploration of the experience of taking care of the suffering adolescents.

SUMMARY:
The purpose of this study is to explore the perspectives of health professionals on chronic (non-malignant) musculoskeletal pain in adolescence and young adulthood. The prevalence of this pain symptom is rising for ten years, and most of the time the diagnosis is complex. Health professionals have to differentiate between the continuing activity of a somatic problem, some painful sequelae, a low threshold for the perception of pain, and psychological symptoms with somatic expression. Diagnosis in this case takes time, and is a matter of trained specialists. No protocol exists to assess the sub-clinical symptoms which will be used to help doing this complex task.

This qualitative study will elicit the perspectives of trained specialists on this diagnosis: how do they deal with these patients? What signs and symptoms helps them? The results will present their clinical experiences. The overall goal is to construct the first chronic musculoskeletal pain multidimensional scale that will help the practitioners with this complex diagnosis.

DETAILED DESCRIPTION:
Recent research suggests that musculoskeletal pain may be the most common complaint for which children are referred to a pediatric rheumatologist and is present in approximately 50% of all new patients. A small percentage of these patients will be diagnosed with a form of juvenile idiopathic arthritis (JIA), which is marked by clinically significant pain. A larger percentage will be diagnosed with a musculoskeletal pain syndrome, that approximately 25% of them are chronic and defined as > = 3 months. The chronic pain symptom is a subjective one that professionals have to precise its outlines in term of semiology, nature and efficacity of past treatments, medical and family backgrounds. The professional then will have to pinpoint a diagnosis, while assessing the consequences of the pain and treating it.

Most of the time this task is a complex one and professionals have to build their diagnostic on a body of clinical, paraclinical and more social, familial and psychological evidences. No clear protocol exists to help the professionals with differentiating the continuing activity of a somatic problem, some painful sequelae, a low threshold for the perception of pain, and psychological symptoms with somatic expression. This diagnostic process is lying on sub-clinical symptoms that investigators have to elicit in order to help professionals to better support their patients.

This qualitative study will explore the daily clinical experience of the health professionals involved in the care of adolescents suffering from chronic musculoskeletal pain. Semi-structured interviews will be analyzed with a phenomenological approach (interpretative phenomenological analysis). The rich phenomenological description will be the first step of a more ambitious project of constructing a multidimensional scale that will help the practitioners with this complex diagnosis.

ELIGIBILITY:
Inclusion Criteria:

* Health care professionals working with the French National Reference in Center Pediatric Rheumatology and Inflammatory Diseases
* Professional experiences on the care of chronic musculoskeletal pain

Exclusion Criteria:

- Refusal to participate in the study

Ages: 25 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study will concern the health professionals who takes care of adolescents suffering from chronic (non-malignant) musculoskeletal pain. In France, the medical specialities concerned are paediatric medicine, rheumatology, pain medicine, adolescent medicine and psychiatry. The investigators also want to include participants from paramedical fields: physiotherapists, ergotherapists and psychologists. The participants will be selected in the large repository of the professionals working with the French National Reference Center in Paediatric Rheumatology and Inflammatory Diseases
Sampling Method: Non-Probability Sample
Enrollment: 25 (Actual)
Dates: Start 2017-09-21 (Actual); Primary Completion 2018-01-30 (Actual); Study Completion 2018-01-30 (Actual)

PRIMARY OUTCOMES:
Qualitative description of the experience of health professionals faced to adolescents consulting for chronic (non-malignant) musculoskeletal pain | 1 day
  The data collection will consist in health professionals' interviews. All the content of the interviews will be included in the data analysis. The interviews will contain the deepest experience of these professionals in their confrontation of adolescents who present chronic musculoskeletal pain.

CONTACTS AND LOCATIONS:
Overall Officials: Pierre QUARTIER, MD, PhD, Study Chair — Assistance Publique - Hôpitaux de Paris; Jonathan LACHAL, MD, PhD, Study Chair — Assistance Publique - Hôpitaux de Paris
Locations (2):
- France (2):
  - Cochin hospital, Paris, Paris
  - Necker Hospital, Paris, Paris

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Goodman JE, McGrath PJ. The epidemiology of pain in children and adolescents: a review. Pain. 1991 Sep;46(3):247-264. doi: 10.1016/0304-3959(91)90108-A. No abstract available. PMID 1758709
- [Background] De Inocencio J. Epidemiology of musculoskeletal pain in primary care. Arch Dis Child. 2004 May;89(5):431-4. doi: 10.1136/adc.2003.028860. PMID 15102634
- [Background] Anthony KK, Schanberg LE. Pediatric pain syndromes and management of pain in children and adolescents with rheumatic disease. Pediatr Clin North Am. 2005 Apr;52(2):611-39, vii. doi: 10.1016/j.pcl.2005.01.003. PMID 15820381
- [Background] Petty RE, Southwood TR, Manners P, Baum J, Glass DN, Goldenberg J, He X, Maldonado-Cocco J, Orozco-Alcala J, Prieur AM, Suarez-Almazor ME, Woo P; International League of Associations for Rheumatology. International League of Associations for Rheumatology classification of juvenile idiopathic arthritis: second revision, Edmonton, 2001. J Rheumatol. 2004 Feb;31(2):390-2. No abstract available. PMID 14760812
- [Background] Jaremko JL, Liu L, Winn NJ, Ellsworth JE, Lambert RG. Diagnostic utility of magnetic resonance imaging and radiography in juvenile spondyloarthritis: evaluation of the sacroiliac joints in controls and affected subjects. J Rheumatol. 2014 May;41(5):963-70. doi: 10.3899/jrheum.131064. Epub 2014 Mar 15. PMID 24634199
- [Background] Bell DS, Bell KM, Cheney PR. Primary juvenile fibromyalgia syndrome and chronic fatigue syndrome in adolescents. Clin Infect Dis. 1994 Jan;18 Suppl 1:S21-3. doi: 10.1093/clinids/18.supplement_1.s21. PMID 8148447
- [Background] McGhee JL, Burks FN, Sheckels JL, Jarvis JN. Identifying children with chronic arthritis based on chief complaints: absence of predictive value for musculoskeletal pain as an indicator of rheumatic disease in children. Pediatrics. 2002 Aug;110(2 Pt 1):354-9. doi: 10.1542/peds.110.2.354. PMID 12165590
- [Background] Sherry DD, McGuire T, Mellins E, Salmonson K, Wallace CA, Nepom B. Psychosomatic musculoskeletal pain in childhood: clinical and psychological analyses of 100 children. Pediatrics. 1991 Dec;88(6):1093-9. PMID 1956724
- [Background] Kashikar-Zuck S, Goldschneider KR, Powers SW, Vaught MH, Hershey AD. Depression and functional disability in chronic pediatric pain. Clin J Pain. 2001 Dec;17(4):341-9. doi: 10.1097/00002508-200112000-00009. PMID 11783815
- [Background] - Lachal J, Speranza M, Schmitt A, Spodenkiewicz M, Falissard B, Moro MR, Revah-Levy A. Depression in adolescent from qualitative research to measurement. Adolescent Psychiatry 2012,2(4):296-308.
- [Background] - Smith J. Interpretative phenomenological analysis. In: Qualitative Psychology: A Practical Guide to Research Methods. 2e éd. Sage Publications Ltd; 2008.
- [Background] Taieb O, Bricou O, Baubet T, Gaboulaud V, Gal B, Mouthon L, Dhote R, Guillevin L, Rose Moro M. Patients' beliefs about the causes of systemic lupus erythematosus. Rheumatology (Oxford). 2010 Mar;49(3):592-9. doi: 10.1093/rheumatology/kep430. Epub 2009 Dec 29. PMID 20040529
- [Background] Smith JA, Michie S, Stephenson M, Quarrell O. Risk Perception and Decision-making Processes in Candidates for Genetic Testing for Huntington's Disease: An Interpretative Phenomenological Analysis. J Health Psychol. 2002 Mar;7(2):131-44. doi: 10.1177/1359105302007002398. PMID 22114233
- [Background] Chapman E, Smith JA. Interpretative phenomenological analysis and the new genetics. J Health Psychol. 2002 Mar;7(2):125-30. doi: 10.1177/1359105302007002397. PMID 22114232
- [Result] Lefevre H, Loisel A, Meunier BB, Deslandre C, Lemoine N, Moro MR, Quartier P, Lachal J. Chronic idiopathic musculoskeletal pain in youth: a qualitative study. Pediatr Rheumatol Online J. 2019 Dec 27;17(1):86. doi: 10.1186/s12969-019-0389-3. PMID 31882011
- See also: QSR International. Logiciel NVivo pour la recherche qualitative - de l'analyse de contenu et de l'évaluation jusqu'à l'étude de marché [Internet]. 2015 [cité 30 juill 2015] — http://www.qsrinternational.com/other